CLINICAL TRIAL: NCT01366586
Title: Confocal Laser Endomicroscopy for in Vivo Molecular Imaging of Gastric Cancer by Targeting MG7 Antigen
Brief Title: Confocal Laser Endomicroscopy for in Vivo Molecular Imaging of Gastric Cancer by Targeting MG7-Ag
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Chief of the Department of Gastroenterology, Qilu Hospital, Shandong University, Shandong University
Other Study IDs: 2011SDU-QILU-G02
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Taken biopsies during endoscopy
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study aims to:

1. Achieve molecular imaging of MG7 antigen in patients with gastric cancer in vivo using confocal laser endomicroscopy.
2. Compare the results of in vivo MG7-specific molecular imaging with CLE and ex vivo immunohistochemistry .

DETAILED DESCRIPTION:
Gastric cancer remains the world's second leading cause of cancer-related death. Improved prognosis essentially depend on earlier diagnosis. Gastric monoclonal antibody MG7 has been validated as a specific antibody in gastric cancerous tissue. Conventional evaluation of MG7 antigen expression is immunohistochemistry, which is time-consuming, and the immunoreactivity can be affected by storage and fixation of tissue. Confocal laser endomicrosopy enables visualization of the cellular and subcellular structures in vivo. Thus this study aims to achieve molecular imaging of MG7 antigen in gastric cancer in vivo using confocal laser endomicroscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients with endoscopically diagnosed gastric cancer

Exclusion Criteria:

* Patients who are allergic to fluorescein sodium
* Patients who are unwilling to sign or give the informed consent form
* Patients with giant tumors or obvious GI tract bleeding which make it hard or impossible to observe the lesions
* Patients with impaired cardiac, liver or renal function
* Patients with coagulopathy
* Patients with pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with endoscopically diagnosed gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD, PhD, Study Director — Department of Gastroenterology, Qilu Hospital
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China